CLINICAL TRIAL: NCT03937154
Title: PROCLAIM: A Phase 3 Randomized Placebo-controlled Double-blind Study of Romiplostim for the Treatment of Chemotherapy-induced Thrombocytopenia in Patients Receiving Chemotherapy for Treatment of Non-small Cell Lung Cancer (NSCLC), Ovarian Cancer, or Breast Cancer
Brief Title: Study of Romiplostim for Chemotherapy-induced Thrombocytopenia in Adult Subjects With Non-small Cell Lung Cancer (NSCLC), Ovarian Cancer, or Breast Cancer
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20170770
Record Dates: First submitted 2019-04-24; First posted 2019-05-03 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Chemotherapy-induced Thrombocytopenia
Keywords: Chemotherapy-induced thrombocytopenia; Non-small Cell Lung Cancer; Ovarian Cancer; Breast Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Ovarian Neoplasms; Breast Neoplasms | interventions — romiplostim

STUDY DESIGN:
Intervention Model Description: The study will consist of a screening period of up to 4 weeks, a treatment period long enough to allow for assessment of 3 planned cycles of chemotherapy, a follow-up visit, and LTFU. Given that subjects are required to have 3 remaining planned cycles of chemotherapy, the chemotherapy cycles may be 3 or 4 weeks in duration, and the investigational product dose adjustment guidelines allow for up to 12 weeks of dosing before a subject is declared a non-responder, the majority of study subjects will receive investigational product for a range of 10-24 weeks.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Romiplostim (Experimental): The study in a 2:1 randomization ratio(108 subjects to romiplostim). Amgen investigational product (romiplostim or placebo) will be administered in the clinic by a qualified healthcare provider as a subcutaneous injection.
  Interventions: Drug: Romiplostim
- Placebo (Placebo Comparator): The study in a 2:1 randomization ratio (54 subjects to placebo) Amgen investigational product (romiplostim or placebo) will be administered in the clinic by a qualified healthcare provider as a subcutaneous injection.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Romiplostim — This study is designed to study Romiplostim for the treatment of chemotherapy-induced thrombocytopenia (CIT) in patients receiving chemotherapy for the treatment of non-small cell lung cancer (NSCLC), ovarian cancer, or breast cancer
  Other Names: Nplate
  Arms: Romiplostim
Drug: Placebo — Placebo comparator
  Arms: Placebo

SUMMARY:
To evaluate the efficacy of romiplostim for the treatment of CIT in patients receiving chemotherapy for the treatment of NSCLC, ovarian cancer, or breast cancer measured by the ability to administer on-time, full-dose chemotherapy

DETAILED DESCRIPTION:
This is a phase 3, randomized, placebo-controlled, multicenter, international study for the treatment of CIT in adult subjects receiving chemotherapy for the treatment of NSCLC, ovarian cancer, or breast cancer. Subjects must have a platelet count ≤ 85 x 10^9/L on day 1 of the study. The study will consist of a screening period of up to 4 weeks, a treatment period long enough to allow for assessment of 3 planned cycles of chemotherapy, a follow-up visit, and long-term follow-up (LTFU). Given that subjects are required to have 3 remaining planned cycles of chemotherapy, the chemotherapy cycles may be 3 or 4 weeks in duration, and the investigational product dose adjustment guidelines allow for up to 12 weeks of dosing before a subject is declared a non-responder, the majority of study subjects will receive investigational product for a range of 10-24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Subject has provided informed consent prior to initiation of any study-specific activities/procedures or subject's legally acceptable representative has provided informed consent prior to any study-specific activities/procedures being initiated when the subject has any kind of condition that, in the opinion of the investigator, may compromise the ability of the subject to give written informed consent.
* Males or females greater than or equal to 18 years of age at signing of the informed consent.
* Documented active stage I, II, III or IV locally advanced or metastatic of the following tumor types: NSCLC, breast cancer, or ovarian cancer (includes fallopian tube epithelial carcinomas and peritoneal epithelial carcinoma of unknown primary), or any stage recurrent disease. Patients with documented locally advanced (stage III) NSCLC should not be amenable to definitive treatment with chemoradiation and/or surgery.
* Subjects must be receiving cancer treatment with 21- or 28-day cycles, using one of the following carboplatinum-based combination chemotherapy regimens: carboplatin/gemcitabine based, carboplatin/pemetrexed based, carboplatin/liposomal doxorubicin based or carboplatin/taxane based (which includes either paclitaxel, nab-paclitaxel, or docetaxel) or single agent chemotherapy regimen with any of the above mentioned drugs. Use of combination regimens with one of the above carboplatinum-based regimens is permitted with (1) anti-angiogenic agents (such as bevacizumab); (2) targeted therapy (such as anti-epidermal growth factor agents or anti- human epidermal growth factor receptor 2) or (3) immune checkpoint inhibitors. Cycle duration is based on intervals between day 1 of chemotherapy cycles (overlapping with carboplatin intervals) every 21 or 28 day cycles for single agent regimens. OR, Subjects must have CIT from a non-protocol chemotherapy regimen, planning to start treatment with one of the above protocol chemotherapy regimens which has been delayed ≥ 1 week due to CIT.
* Subjects must have a local platelet count ≤ 85 x 109/L on day 1 of the study.
* Subjects must be at least 21 or 28 days removed from the start of the chemotherapy cycle immediately prior to study day 1 if receiving a 21-day or 28-day cycle chemotherapy regimen, respectively.
* Subjects must have at least 3 remaining planned cycles of chemotherapy at study enrollment.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2.

Exclusion Criteria:

* Acute lymphoblastic leukemia.
* Acute myeloid leukemia.
* Any myeloid malignancy.
* Myelodysplastic syndrome. Baseline bone marrow biopsy is not required to rule out MDS. However, if a bone marrow biopsy and cytogenetics were performed as part of diagnostic or staging work-up, these results will be collected to confirm.
* Myeloproliferative disease.
* Multiple myeloma.
* Within 4 months prior to enrollment, any history of active congestive heart failure (New York Heart Association [NYHA] Class III to IV), symptomatic ischemia, uncontrolled arrhythmias, clinically significant electrocardiogram (ECG) abnormalities, screening ECG with corrected QT (QTc) interval of greater than 470 msec, pericardial disease, or myocardial infarction.
* Major surgery less than or equal to 28 days or minor surgery less than or equal to 3 days prior to enrollment.
* New or uncontrolled venous thromboembolism or thrombotic events within 3 months prior to screening. To be eligible, subjects must have received at least 14 days of anticoagulation for a new thrombotic event and considered to be stable and suitable for continued therapeutic anticoagulation during trial participation.
* History of arterial thrombotic events (eg, myocardial ischemia, transient ischemic attack, or stroke) within 6 months prior to screening.
* Evidence of active infection within 2 weeks prior to the first dose of study treatment.
* Known human immunodeficiency virus infection with any detectable viral load at screening. Subjects without a documented diagnosis in their medical history will require a local laboratory assessment at screening. If local laboratory results are not available use central laboratory results.
* Known active of chronic hepatitis C or hepatitis B infection. Subjects without a documented diagnosis in their medical history will require a local laboratory assessment at screening. If local laboratory results are not available use central laboratory results. Hepatitis B and C infection is based on the following results:
* Positive for hepatitis B surface antigen (HBsAg) (indicative of chronic hepatitis B or recent acute hepatitis B).
* Negative HBsAg and positive for hepatitis B core antibody: hepatitis B virus DNA by polymerase chain reaction (PCR) is necessary. Detectable hepatitis B virus DNA suggests occult hepatitis B.
* Positive hepatitis C virus antibody: hepatitis C virus RNA by PCR is necessary. Detectable hepatitis C virus RNA suggests chronic hepatitis C.
* In addition to the conditions listed in exclusion criteria 201 through 206, secondary malignancy within the past 5 years except:
* Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease.
* Adequately treated cervical carcinoma in situ without evidence of disease.
* Adequately treated breast ductal carcinoma in situ without evidence of disease.
* Prostatic intraepithelial neoplasia without evidence of prostate cancer.
* Adequately treated urothelial papillary noninvasive carcinoma or carcinoma in situ.
* Malignancy treated with curative intent and with no known active disease present for greater than or equal to 3 years before enrollment and felt to be at low risk for recurrence by the treating physician (excluding malignancies listed in exclusion criteria 201 - 206).
* Thrombocytopenia due to another etiology other than CIT (eg, chronic liver disease, prior history of immune thrombocytopenia purpura).
* Any combined modality regimen containing radiation therapy or surgery occurring concomitantly with neo-adjuvant chemotherapy or where radiation therapy is planned during the cycle preceding 3 planned on-study cycles of chemotherapy.

Prior/Concomitant Therapy:

- Previous use of romiplostim, pegylated recombinant human megakaryocyte growth and development factor, eltrombopag, recombinant human TPO, any other TPO receptor agonist, or any investigational platelet producing agent.

Prior/Concurrent Clinical Study Experience - Currently receiving (or plan to receive) treatment in another investigational device or drug study, or less than 28 days since ending treatment on another investigational device or drug study(ies). Other investigational procedures while participating in this study are excluded.

Diagnostic Assessments

* Anemia (hemoglobin < 80 g/L [8 g/dL]) on the day of initiation of investigational product as assessed by local labs. Use of red cell transfusions and erythropoietic stimulating agents is permitted throughout the study as per institutional guidelines.
* Neutropenia (absolute neutrophil count less than 1 x 10 9/L) on the day of initiation of investigational product as assessed by local labs. Use of granulocyte-colony stimulating factor is permitted throughout the study as per institutional guidelines.
* Abnormal renal function with creatinine clearance less than 30 mL/min using the Cockcroft-Gault estimated creatinine clearance as assessed by local laboratory. If local laboratory results are not available use central laboratory results.

during screening.

- Abnormal liver function (total bilirubin greater than 3X ULN; alanine aminotransferase [ALT] or aspartate aminotransferase [AST] greater than 3X ULN for subjects without liver metastases or greater than or equal to 5X ULN for subjects with liver metastases) as assessed by local laboratory during screening. If local laboratory results are not available use central laboratory results.

Other Exclusions

* Females who are pregnant or breastfeeding or planning to become pregnant or breastfeed during treatment and for an additional 7 months after treatment (and chemotherapy) discontinuation (females of childbearing potential should only be included after a confirmed menstrual period and a negative highly sensitive urine or serum pregnancy test.)
* Females of childbearing potential unwilling to use a highly effective method of contraception during treatment and for an additional 7 months after treatment (and chemotherapy) discontinuation. Refer to Appendix 5 for additional contraceptive information.
* Males unwilling to use contraception* (male condom or sexual abstinence) or their female partner(s) of childbearing potential who are unwilling to use a highly effective method of contraception during treatment (and chemotherapy) and for an additional 7 months after treatment (and chemotherapy) discontinuation. *If the male's sole partner is of non-childbearing potential, he is not required to use additional forms of contraception during the study.
* Subject has known sensitivity to any of the products to be administered during dosing.
* Subject likely to not be available to complete all protocol-required study visits or procedures, and/or to comply with all required study procedures (eg, COAs) to the best of the subject and investigator's knowledge.
* History or evidence of any other clinically significant disorder, condition or disease (with the exception of those outlined above) that, in the opinion of the investigator or Amgen physician, if consulted, would pose a risk to subject safety or interfere with the study evaluation, procedures or completion.
* Male subjects with a pregnant partner who are unwilling to practice abstinence or use a condom during treatment (and chemotherapy) and for an additional 7 months after treatment (and chemotherapy) discontinuation.
* Male subjects unwilling to abstain from donating sperm during treatment (and chemotherapy) and for an additional 7 months after treatment (and chemotherapy) discontinuation.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2020-02-26 (Actual); Primary Completion 2026-05-20 (Estimated); Study Completion 2027-05-20 (Estimated)

PRIMARY OUTCOMES:
Incidence of either a chemotherapy dose delay or reduction | 48 days
  No thrombocytopenia-induced modification of any myelosuppressive agent in the second and third cycles of the planned on-study chemotherapy regimen. Thrombocytopenia-induced modifications include chemotherapy dose reduction, delay, omission, or chemotherapy treatment discontinuation due to platelet counts below 100 x 109/L

SECONDARY OUTCOMES:
Depth of Platelet Count | 48 days
  the depth of the platelet count nadir from the start of the first on-study chemotherapy cycle through the end of the treatment period
Time to First platelet response | 7 days
  The time to first platelet response, defined by platelet count ≥ 100 x 109/L in the absence of platelet transfusions during the preceding 7 days
the duration-adjusted event rate of ≥ grade 2 bleeding events | 48 days
  the duration-adjusted event rate of ≥ grade 2 bleeding events, as assessed by Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 grading scale
Overall survival | 1 Year
  1-year overall survival
Proportion of subjects with at leat 1 incidence of platelet transfusion | 48 days
  platelet transfusion(s) during the treatment period
proportion of patients achieving platelet count >= 100 x 10 9/L | 7 days
  7 days after 3rd dose of IP with no transfusions in preceding 7 days
The subject incidence of adverse events | 36 months
  Through end of study, up to 36 months. It will be counted in as an adverse event: any treatment - emergent adverse events, fatal adverse events, serious adverse events, or clinically significant changes in laboratory values.
Number of subjects who develop anti-romiplostim antibodies | 36 Months
  Through end of study up to 36 months
Number of subjects who develop anti-TPO antibodies | 36 months
  Through end of study, up to 36 months
Number of subjects who experience myelodysplastic syndromes | 36 months
  Through end of study, up to 36 months
Number of subjects who experience secondary malignancies | 36 months
  Through end of study, up to 36 months

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (138):
- United States (27):
  - Saint Bernards Medical Center, Jonesboro, Arkansas
  - Los Angeles Cancer Network, Anaheim, California
  - University of California Irvine, Orange, California
  - Colorado West Healthcare System dba Grand Valley Oncology, Grand Junction, Colorado
  - University of Miami School of Medicine, Miami, Florida
  - Ocala Oncology Center, Ocala, Florida
  - Mid Florida Hematology and Oncology Centers PA, Orange City, Florida
  - Saint Alphonsus Regional Medical Center, Boise, Idaho
  - University of Chicago, Chicago, Illinois
  - Orchard Healthcare Research Inc, Skokie, Illinois
  - Christus Saint Frances Cabrini Hospital, Alexandria, Louisiana
  - University Medical Center New Orleans, New Orleans, Louisiana
  - Christus Highland Cancer Treatment Center, Shreveport, Louisiana
  - Mercy Medical Center, Baltimore, Maryland
  - American Oncology Partners, PA, Bethesda, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Hattiesburg Clinic Hematology/Oncology, Hattiesburg, Mississippi
  - Oncology Hematology Associates, Springfield, Missouri
  - Great Falls Clinic, Great Falls, Montana
  - Nebraska Cancer Specialists, Omaha, Nebraska
  - Regional Cancer Care Associates, Sparta, New Jersey
  - Broome Oncology LLC, Binghamton, New York
  - Saint Lukes University Health Network, Bethlehem, Pennsylvania
  - The Center for Cancer and Blood Disorders, Fort Worth, Texas
  - Community Cancer Trials of Utah, Ogden, Utah
  - Medical Oncology Associates PS, Spokane, Washington
  - Yakima Valley Memorial Hospital, Yakima, Washington
- Argentina (4):
  - Instituto Oncologico Cordoba, Córdoba, Córdoba Province
  - Centro Medico Austral, Buenos Aires, Distrito Federal
  - Centro de Investigaciones Clínicas Clínica Viedma, Viedma, Río Negro Province
  - Centro de Diagnostico Investigacion y Tratamiento, Salta
- Medizinische Universitaet Innsbruck, Innsbruck, Austria
- Brazil (11):
  - Instituto de Oncologia do Parana, Curitba, Paraná
  - Vencer e Oncoclinica, Teresina, Piauí
  - Liga Norte-Riograndense Contra O Cancer, Natal, Rio Grande do Norte
  - Centro de Pesquisa da Serra Gaucha - Cepesg, Caxias do Sul, Rio Grande do Sul
  - Associação Hospitalar Moinhos de Vento, Porto Alegre, Rio Grande do Sul
  - Clinica de Neoplasias Litoral, Itajaí, Santa Catarina
  - Hospital de Amor, Barretos, São Paulo
  - Loema Instituto de Pesquisa Clinica e Consultores Ltda - Clinica Loema, Campinas, São Paulo
  - Hospital de Base de Sao Jose do Rio Preto, São José do Rio Preto, São Paulo
  - Casa de Saude Santa Marcelina, São Paulo, São Paulo
  - Pérola Clínica de Pesquisa e Centro de Estudos em Oncologia Ginecológica e Mamaria Ltda, São Paulo
- Bulgaria (3):
  - Complex Oncology Center - Ruse EOOD, Rousse
  - Multiprofile Hospital for Active Treatment Serdika EOOD, Sofia
  - Specialized Hospital for Active Treatment of Oncology EAD, Sofia
- Chile (2):
  - James Lind Centro de Investigacion del Cancer, Temuco, Cautín
  - Orlandi Oncologia, Santiago
- Colombia (2):
  - Oncomedica Imat, Montería, Departamento de Córdoba
  - Centro Medico Imbanaco, Cali, Valle del Cauca Department
- Greece (9):
  - Agios Savvas Anticancer Hospital, Athens
  - Henry Dunant Hospital Center, Athens
  - Sotiria General Hospital, Athens
  - Alexandra Hospital, Athens
  - Attikon University Hospital, Athens
  - University Hospital of Heraklion, Heraklion - Crete
  - Metaxa Anticancer Hospital, Piraeus
  - Agios Loukas Clinic, Thessaloniki
  - Iatriko Diavalkaniko Thessalonikis, Thessaloniki
- Hungary (6):
  - Semmelweis Egyetem, Budapest
  - Farkasgyepui Tudogyogyintezet, Farkasgyepű
  - Gyor-Moson-Sopron Varmegyei Petz Aladar Egyetemi Oktatokorhaz, Győr
  - Fejer Varmegyei Szent Gyorgy Egyetemi Oktato Korhaz, Székesfehérvár
  - Jasz-Nagykun-Szolnok Varmegyei Hetenyi Geza Korhaz-Rendelointezet, Szolnok
  - Reformatus Pulmonologiai Centrum, Törökbálint
- Mexico (6):
  - Oncotech, La Paz, Baja California Sur
  - Centro de Atencion e Investigacion Cardiovascular del Potosi Sc, San Luis Potosí City, San Luis Potosí
  - Phylasis Clinical Research, Cuautitlán Izcalli
  - Centro Medico Nacional Siglo XXI, México
  - Oaxaca Site Management Organization SC, Oaxaca City
  - Phylasis Clinicas Research Toluca, Toluca
- Peru (2):
  - Hospital Goyeneche, Arequipa
  - Oncosalud, Lima
- Poland (10):
  - Powiatowe Centrum Zdrowia w Brzezinach Sp Z o o, Brzeziny
  - Centrum Onkologii im prof Franciszka Lukaszczyka w Bydgoszczy, Bydgoszcz
  - Szpital Wojewodzki imienia Mikolaja Kopernika w Koszalinie, Koszalin
  - Centrum Onkologii Ziemi Lubelskiej im sw Jana z Dukli, Lublin
  - Uniwersytecki Szpital Kliniczny w Poznaniu, Poznan
  - Wojewodzki Szpital im Sw Ojca Pio w Przemyslu, Przemyśl
  - Uniwersytecki Szpital Kliniczny nr 2 Pum w Szczecinie, Szczecin
  - Provita Centrum Medyczne Spzoo, Tomaszów Mazowiecki
  - Specjalistyczny Szpital im Dra Alfreda Sokolowskiego, Wałbrzych
  - Dolnoslaskie Centrum Onkologii, Pulmonologii i Hematologii, Wroclaw
- Portugal (4):
  - Unidade Local de Saude de Santa Maria, EPE - Hospital Pulido Valente, Lisbon
  - Unidade Local de Saude de Matosinhos, EPE - Hospital Pedro Hispano, Matosinhos Municipality
  - Unidade Local de Saude de Santo Antonio, EPE - Hospital de Santo Antonio, Porto
  - Unidade Local de Saude de Sao Joao, EPE - Hospital de Sao Joao, Porto
- Romania (10):
  - Spitalul Universitar de Urgenta Elias, Bucharest
  - Memorial Healthcare International SRL, Bucharest
  - Institutul Oncologic, Prof Dr Alexandru Trestioreanu, Bucharest
  - Spitalul Clinic Coltea, Bucharest
  - Institutul Oncologic Prof Dr Ion Chiricuta Cluj-Napoca, Cluj-Napoca
  - SC Medisprof SRL, Cluj-Napoca
  - Oncolab, Craiova
  - Institutul Regional de Oncologie Iasi, Iași
  - Spitalul Municipal Ploiesti, Ploieşti
  - SC Oncomed SRL, Timișoara
- Russia (12):
  - SBHI of Arkhangelsk region Arkhangelsk clinical oncology dispensary, Arkhangelsk
  - Autonomic SHI Republican clinical oncology dispensary of MoH of the Republic of Tatarstan, Kazan'
  - State Healthcare Institution Goroda Moskvi City Clinical Hospital 1, Moscow
  - Clinical hospital 2, Group of companies medsi, Moscow
  - Medsi Group, Moscow Region
  - LLC Tonus, Nizhny Novgorod
  - Omsk Regional Clinical Oncology Dispensary, Omsk
  - State budget institution of public health Pyatigorsk oncology dispensary, Pyatigorsk
  - State Institution of Public Health, Ryazan
  - State Institution of Public Health Oncology Dispensary 2 of Public Health Krasnodar Region, Sochi
  - State Institution of Public Health Tambov Regional Oncology Dispensary, Tambov
  - Respublican clinical oncology dispensary Minzdrava of Republic of Bashkortostan, Ufa
- Spain (9):
  - Hospital Clinico Universitario San Cecilio, Granada, Andalusia
  - Hospital Universitario Nuestra Señora de Valme, Seville, Andalusia
  - Hospital Universitario Virgen del Rocio, Seville, Andalusia
  - Hospital Clinico Universitario de Salamanca, Salamanca, Castille and León
  - Instituto Oncologico IOB, Barcelona, Catalonia
  - Hospital Santa Maria Nai, Ourense, Galicia
  - Hospital Universitario de Fuenlabrada, Fuenlabrada, Madrid
  - Consorcio Hospitalario Provincial de Castellon, Castellon, Valencia
  - Hospital Universitario Madrid Sanchinarro, Madrid
- Turkey (Türkiye) (17):
  - Saglik Bilimleri Universitesi Gulhane Egitim ve Arastirma Hastanesi, Ankara
  - Doktor Abdurrahman Yurtaslan Ankara Onkoloji Egitim ve Arastirma Hastanesi, Ankara
  - Saglik Bilimleri University Ankara Ataturk Chest Diseases and Chest Surgery Training and Research Ho, Ankara
  - Memorial Ankara Hastanesi, Ankara
  - Ankara Bilkent Sehir Hastanesi, Ankara
  - Pamukkale Universitesi Tip Fakultesi Hastanesi, Denizli
  - Trakya Universitesi Saglik Arastirma ve Uygulama Merkezi, Edirne
  - Istanbul Universitesi Cerrahpasa Tip Fakultesi, Istanbul
  - Basaksehir Cam ve Sakura Sehir Hastanesi, Istanbul
  - Marmara Universitesi Tip Fakultesi Hastanesi, Istanbul
  - Izmir Katip Celebi Universitesi Ataturk Egitim ve Arastirma Hastanesi, Izmir
  - Izmir Ekonomi Universitesi Medical Point Hastanesi, Izmir
  - Kocaeli Universitesi Tip Fakultesi Hastanesi, Kocaeli
  - Necmettin Erbakan Universitesi Tip Fakultesi Hastanesi, Konya
  - Inonu Universitesi Turgut Ozal Tip Merkezi, Malatya
  - Sakarya Egitim ve Arastirma Hastanesi, Sakarya
  - Namik Kemal Universitesi Hastanesi, Tekirdağ
- Ukraine (3):
  - Communal Institution Chernivtsi Regional Clinical Oncological Dispensary, Chernivtsi
  - Transcarpathian Regional Clinical Oncological Dispensary, Uzhhorod
  - Vinnytsya Regional Clinical Oncological Dispensary, Vinnytsia

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication (or other new use) have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors, and if not approved, may be further arbitrated by a Data Sharing Independent Review Panel. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: https://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com